CLINICAL TRIAL: NCT05855174
Title: Protein and Exercise-Induced Gastrointestinal Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mount Royal University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: MountRoyalU
Record Dates: First submitted 2023-03-22; First posted 2023-05-11 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: Gastro-Intestinal Disorder
Keywords: Dietary protein; Runners; Gastrointestinal symptoms
MeSH Terms: conditions — Digestive System Diseases | interventions — Whey Proteins

STUDY DESIGN:
Intervention Model Description: Crossover intervention; all participants will have a low protein and a high protein session.
Who Masked: Participant
Masking Description: In this single-blinded crossover design, the participants will be blinded to which intervention the participants are receiving (i.e., high protein or low protein drinks).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low Protein (Active Comparator): Protein intake at 0.15g/kg body weight
  Interventions: Dietary Supplement: Whey protein
- High Protein (Experimental): Protein intake at 0.4 g/kg body weight
  Interventions: Dietary Supplement: Whey protein

INTERVENTIONS:
Dietary Supplement: Whey protein — Weight protein provided in a shake with carbohydrate and water

SUMMARY:
Recommendations for carbohydrate intakes in the pre-exercise meal for endurance athletes are available; however, are lacking protein. Therefore, the purpose of this study is to quantify exercise-induced gastrointestinal symptoms and gut fullness occurring in response to a low protein (control) and a high protein (intervention) pre-exercise meal. The secondary purpose is to quantify blood glucose responses to a high-protein pre-exercise meal as compared to a low-protein control.

DETAILED DESCRIPTION:
Context: Proper nutrition is crucial for peak sport performance. Recommendations for carbohydrate intakes in the pre-exercise meal for endurance athletes are available; however, are lacking for protein. Furthermore, a recent position statement regarding nutrient timing for exercise also lacks protein recommendations. The only advice provided is to avoid "too much" as it may cause gastrointestinal (GI) discomfort. The aforementioned recommendation provides no guidance as to how much is "too much" nor, to our knowledge, is there any clinical trial data to support the position. Exercise-associated gastrointestinal symptoms are a common cause of withdrawal from competition; thus, athletes need to consider the impact of dietary choices on gastrointestinal (GI) symptoms, as well as performance. Exercise induced GI symptoms can plague all athletes; but the effects seem to be most pronounced in endurance running. The reported prevalence of exercise-induced GI disturbances varies depending on methodology; however a questionnaire administered by the investigator's lab to 440 runners found 41% experienced stomach pain/cramps, 24% had intestinal issues, and over 20% reported bloating, diarrhea and/or gas. Exercise related GI complaints have been broadly related to diet. Research from the investigator's lab has found that many of the top foods that are avoided pre-running, to reduce GI symptoms, are those classified as high in protein (legumes, meat, poultry, fish, milk). These observations are based on self-reported data from experienced runners, and require testing in a clinical setting.

Objectives: 1) to quantify exercise induced gastrointestinal symptoms and gut fullness occurring in response to a low protein (control) and high protein (intervention) pre-exercise meal. 2) to quantify blood glucose responses to a high protein pre-exercise meal as compared to a low protein control.

Methods: The study is a single blind crossover design. Endurance runners will be ask to standardize their exercise 3-days prior to testing. The participants will be asked to eat a similar meal in the 24-12 hours pre-testing and fast for 12 hours pre-testing. The participants will be assigned to consume a pre-exercise shake with carbohydrate at 0.75g/kg body weight + water at 5ml/kg body weight and either low whey protein control or high whey protein intervention one hour pre-exercise in a randomized fashion. Participants will then complete a 10 km running protocol at 85% of the participant's race pace on a treadmill in an temperature and humidity controlled room. Gastrointestinal symptoms via self-report questionnaire and blood glucose will be measured at fasting, during the one hour digestive period and post-exercise.

ELIGIBILITY:
Inclusion Criteria:

* recreational competitive runners, defined as running at least 25 km per week
* experiences exercise-induced gastrointestinal symptoms while running

Exclusion Criteria:

* individuals with food allergies,
* gastrointestinal disorders (e.g., celiac disease, irritable bowl syndrome, etc.)
* adherence to a special diet
* pregnancy
* pre-existing medical condition that would prevent them from completing the prescribed exercise
* blood-borne illness

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2019-03-13 (Actual); Primary Completion 2023-12-21 (Actual); Study Completion 2023-12-21 (Actual)

PRIMARY OUTCOMES:
Self-report exercise induced gastrointestinal symptoms | 3 hours per session
  Quantify exercise induced gastrointestinal symptoms via a 0-9 point Likert scale questionnaire including 6 questions for upper abdominal problems, 7 questions for lower abdominal problems and 5 systemic problems. Likert scale questions are administered at fasting, pre-exercise and post-exercise. Questionnaires are administered in response to a low protein (control) and a high protein pre-exercise meal.
Gut fullness | 3 hours per session
  Gut fullness measured using a 100mm visual analogue scale anchored by not full at all and very full at fasting 15, 30 and 60 minutes post-meal and post run. Questionnaires are administered in response to a low protein (control) and a high protein pre-exercise meal.

SECONDARY OUTCOMES:
Plasma glucose levels | 3 hours per session
  Quantify blood glucose levels via a finger prick and blood glucose meter in response to a high protein pre-exercise meal as compared to a low protein control at fasting, 30 minutes post meal, 60 minutes post-meal and post 10 km run.
Perceive exertion | 1 hour per session
  Perceived exertion during the 10 km challenge run will be measured via Borg Rating of Perceived Exertion scale post run.

CONTACTS AND LOCATIONS:
Overall Officials: Jill A Parnell, PhD, Principal Investigator — Mount Royal University
Locations (1):
- Mount Royal University, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Briggs MA, Harper LD, McNamee G, Cockburn E, Rumbold PLS, Stevenson EJ, Russell M. The effects of an increased calorie breakfast consumed prior to simulated match-play in Academy soccer players. Eur J Sport Sci. 2017 Aug;17(7):858-866. doi: 10.1080/17461391.2017.1301560. Epub 2017 Mar 21. PMID 28323574
- [Background] Costa RJS, Snipe RMJ, Kitic CM, Gibson PR. Systematic review: exercise-induced gastrointestinal syndrome-implications for health and intestinal disease. Aliment Pharmacol Ther. 2017 Aug;46(3):246-265. doi: 10.1111/apt.14157. Epub 2017 Jun 7. PMID 28589631
- [Background] Kerksick CM, Arent S, Schoenfeld BJ, Stout JR, Campbell B, Wilborn CD, Taylor L, Kalman D, Smith-Ryan AE, Kreider RB, Willoughby D, Arciero PJ, VanDusseldorp TA, Ormsbee MJ, Wildman R, Greenwood M, Ziegenfuss TN, Aragon AA, Antonio J. International society of sports nutrition position stand: nutrient timing. J Int Soc Sports Nutr. 2017 Aug 29;14:33. doi: 10.1186/s12970-017-0189-4. eCollection 2017. PMID 28919842
- [Background] Parnell JA, Wagner-Jones K, Madden RF, Erdman KA. Dietary restrictions in endurance runners to mitigate exercise-induced gastrointestinal symptoms. J Int Soc Sports Nutr. 2020 Jun 10;17(1):32. doi: 10.1186/s12970-020-00361-w. PMID 32522222
- [Background] Pfeiffer B, Stellingwerff T, Hodgson AB, Randell R, Pottgen K, Res P, Jeukendrup AE. Nutritional intake and gastrointestinal problems during competitive endurance events. Med Sci Sports Exerc. 2012 Feb;44(2):344-51. doi: 10.1249/MSS.0b013e31822dc809. PMID 21775906
- [Background] Thomas DT, Erdman KA, Burke LM. Position of the Academy of Nutrition and Dietetics, Dietitians of Canada, and the American College of Sports Medicine: Nutrition and Athletic Performance. J Acad Nutr Diet. 2016 Mar;116(3):501-528. doi: 10.1016/j.jand.2015.12.006. PMID 26920240